CLINICAL TRIAL: NCT04748861
Title: CYCLE-AD: Randomized Controlled Trial to Assess the Efficacy of Indoor Cycling in Slowing Disease Progression in Healthy Older Persons at Genetic Risk for Alzheimer's Disease
Brief Title: CYCLE-AD (CYcling to Cease or Limit the Effects of Alzheimer's Disease)
Acronym: CYCLE-AD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Maryland, College Park (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stephen Rao, Professor, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB20-1198; 1R01AG070736-01 (NIH)
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: High Intensity Exercise; Normal Cognition; Exercise Intervention
Keywords: APOE ε4 allele; indoor cycling; exercise intervention; healthy elders; genetic risk for Alzheimer's Disease

STUDY DESIGN:
Intervention Model Description: A pragmatic, randomized controlled trial with blinded clinical and imaging outcomes
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indoor Cycling (IC) (Experimental): Participants will engage in high-intensity interval training (HIIT; 60-90% of heart rate reserve) in their home via the commercially available Peloton® cycling system or 2) 3x/week (minimum 90 minutes/week) for 18 months.
  Interventions: Other: Indoor Cycling (IC)
- Usual and Customary Care (UCC) (No Intervention): Participants engage in their habitual level of physical activity.

INTERVENTIONS:
Other: Indoor Cycling (IC) — Participants will ride a Peloton bike 3x/week for 18 months.
  Arms: Indoor Cycling (IC)

SUMMARY:
The overall goal of the CYCLE-AD trial is to determine the role of long-term, high intensity exercise in slowing or delaying the onset of cognitive and AD-related brain changes in e4 carriers. Successful translation and demonstration of the effectiveness of a scalable home-based exercise intervention capable of slowing or delaying disease onset will transform AD treatment, improve patient outcomes and quality of life, and reduce health care costs.

DETAILED DESCRIPTION:
The apolipoprotein E epsilon 4 (APOE e4) allele is the most important genetic risk factor for late onset Alzheimer's disease (AD). A recent review by the World Health Organization highlighted the potential protective role of physical activity and exercise against cognitive decline, all-cause dementia, AD, and vascular dementia in healthy individuals. In an 18-month longitudinal observational study, investigators showed that sedentary e4 carriers experience significant declines in episodic memory and hippocampal volume compared to 4 carriers who engaged in moderate PA. Importantly, among 4 non-carriers, no significant longitudinal changes in cognition and brain imaging were observed whether the non-carriers were sedentary or engaged in moderate PA, suggesting that PA has a specific neuroprotective role in delaying the progression of AD in e4 carriers. Based on the results, a pragmatic, randomized controlled trial with blinded clinical and imaging outcomes is proposed to determine the impact of a home based, high intensity exercise intervention in healthy, cognitively intact e4 carriers between the ages of 65 and 80 years. The CYCLE-AD (CYcling to Cease or Limit the Effects of Alzheimer's Disease) trial will recruit otherwise healthy sedentary carriers randomized to one of two groups (n=75 each): 1) an Indoor Cycling (IC) group that participates in high-intensity interval training (HIIT; 60-90% of heart rate reserve) in their home via the commercially available Peloton® cycling system or 2) a Usual and Customary Care (UCC) group, in which participants engage in their habitual level of PA. Investigators hypothesize that an 18-month high-intensity aerobic exercise regimen will slow AD-related disease progression in sedentary elders at genetic risk for AD. Participants in the intervention group will engage in exercise 3x/week (minimum 90 minutes/week) for 18 months. Primary outcome measures, obtained at study entry and at 18 months, will include comprehensive cognitive testing and brain MR imaging to assess disease progression and a comprehensive PA/fitness assessment to measure the degree of change in physical fitness due to high intensity aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy elders, ages 65-80 years, inclusive
2. No cognitive impairment based on screening examination
3. APOE ε4 genotype
4. Inactive; defined as exercising less than 3x per week at moderate-vigorous intensity
5. Fluent in English (a requirement for neurocognitive testing)
6. Does not plan to travel for more than 2 consecutive weeks over the course of the study
7. Demonstrate ability to safely mount and dismount Peloton stationary cycle
8. In-home Wi-Fi (Peloton system requires Wi-Fi to transmit exercise data)
9. Medical clearance by the study doctor to participate in exercise program
10. Participant must meet Peloton height and weight safety requirements

Exclusion Criteria:

1. Any significant neurologic disease, including dementia, mild cognitive impairment, Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, stroke, multiple sclerosis, or history of significant head trauma with a reported loss of consciousness for greater than 30 minutes.
2. Significant medical illnesses/conditions that is unstable and/or uncontrolled (lung or kidney disease, cancer).
3. History of schizophrenia or bipolar disorder.
4. Major Depression within the past year.
5. History of alcohol or substance abuse or dependence within the past 2 years.
6. Current use of Alzheimer's disease medications, including cholinesterase inhibitors and memantine.
7. Any unstable or severe cardiovascular disease or asthmatic condition.
8. History of imaging confirmed transient ischemic attack or a score of >4 on the modified Hachinski ischemic scale.
9. Significant abnormalities in laboratory blood tests that is considered to be a contraindication to exercise.
10. Exclusion criteria specific to MR scanning (weight inappropriate for height, ferrous objects within the body, pregnancy, and a history of claustrophobia).
11. A musculoskeletal issue (arthritis, osteoporosis, back problem) that would limit one's ability to engage in exercise

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning Test Total Recall Trials 1-5 (RAVLT1-5). | 18 months
  Determine the effects of an IC intervention on cognitive functioning
Total Hippocampal Volume (THV) | 18 months
  Determine the effects of an IC intervention on MR brain imaging
V̇O2max | 18 months
  Determine the effects of an IC intervention on PA/fitness testing

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rao, PhD, Principal Investigator — The Cleveland Clinic; Jay Alberts, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States